CLINICAL TRIAL: NCT04997850
Title: The Safety and Efficacy of Transarterial Chemoembolization (TACE) + Lenvatinib +Programmed Cell Death Protein 1 (PD-1) Antibody in the Conversion-resection of Advanced Unresectable Hepatocellular Carcinoma:a Multicenter Prospective Cohort Study
Brief Title: The Safety and Efficacy of Transarterial Chemoembolization (TACE) + Lenvatinib + Programmed Cell Death Protein 1 (PD-1) Antibody of Advanced Unresectable Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xinrui Zhu，MD (Other)
Responsible Party: Sponsor-Investigator, Xinrui Zhu，MD, attending doctor, West China Hospital
Organization: West China Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 311576
Record Dates: First submitted 2021-03-17; First posted 2021-08-10 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Hepatocellular Carcinoma Non-resectable; Transarterial Chemoembolization; Tyrosine Kinase Inhibitor; Immune Checkpoint Blockade
Keywords: Hepatocellular Carcinoma Non-resectable; transarterial chemoembolization; tyrosine kinase inhibitor; immune checkpoint blockade
MeSH Terms: interventions — lenvatinib; camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TACE + lenvastinib + sindilimab/carrelizumab (Experimental): The patients with body weight ≥ 60kg were treated with oral lenvastinib within 3 days (the initial dose was 12mg QD for patients with body weight < 60kg, the initial dose was 8mg QD for patients with body weight < 60kg). After 1-2 weeks of treatment, the patients received the first TACE treatment (3 days before TACE), and continued to take oral lunvastinib 3 days after TACE. Within one week after TACE treatment, 200 mg of sindilimab was given intravenously once every three weeks (every 21 days as a cycle) or 200 mg of carrelizumab was given intravenously once every three weeks (every 21 days as a cycle).
  Interventions: Drug: lenvatinib + sindilimab/carrelizumab; Procedure: TACE
- TACE (Active Comparator): TACE treatment is strictly in accordance with the Chinese guidelines for clinical practice of transcatheter arterial chemoembolization (TACE) for hepatocellular carcinoma (2018 Edition).
  The patients with HCC were selected according to the inclusion criteria (referring to the conditions of the subjects). The subjects who met the inclusion criteria could enter the study after they signed the informed consent. 4-6 weeks after the first TACE treatment, the resectability criteria were evaluated. If not, the next cycle of TACE treatment was carried out. The general principle is to reduce the number of interventional treatment and extend the interval of interventional operation as far as possible under the condition of controlling the tumor and the survival of patients with tumor.
  Interventions: Procedure: TACE

INTERVENTIONS:
Drug: lenvatinib + sindilimab/carrelizumab — 4-6 weeks after the first TACE treatment, the resectability criteria were evaluated. If not, the next treatment cycle was carried out. The trial was terminated if the drug was stopped for more than 28 days due to adverse drug reactions or other reasons. Patients with PD after 6 cycles of sindilimab/carrelizumab treatment were terminated. The follow-up treatment was based on the principle of individualization, multidisciplinary discussion and patients' willingness.
  Arms: TACE + lenvastinib + sindilimab/carrelizumab
Procedure: TACE — TACE treatment is strictly in accordance with the Chinese guidelines for clinical practice of transcatheter arterial chemoembolization (TACE) for hepatocellular carcinoma (2018 Edition).
  The patients with HCC were selected according to the inclusion criteria (referring to the conditions of the subjects). The subjects who met the inclusion criteria could enter the study after they signed the informed consent. 4-6 weeks after the first TACE treatment, the resectability criteria were evaluated. If not, the next cycle of TACE treatment was carried out. The general principle is to reduce the number of interventional treatment and extend the interval of interventional operation as far as possible under the condition of controlling the tumor and the survival of patients with tumor.

SUMMARY:
We adopted the prospective cohort study to compare the safety and efficacy of Transarterial Chemoembolization (TACE) + Lenvatinib + Programmed Cell Death Protein 1 (PD-1) Antibody in the treatment of advanced unresectable liver cancer.The purposes of our study include：1. Primary objective: To compare the safety and efficacy of TACE combined with Lenvatinib and PD-1 antibody versus TACE alone in the conversion-resection of patients with advanced unresectable hepatocellular carcinoma.2. Secondary objective: To compare the long-term outcome of TACE combined with Lenvatinib and PD-1 antibody versus TACE alone for patients with advanced unresectable hepatocellular carcinoma.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (hepatocellular carcinoma,HCC,) accounts for 85% to 90% of primary liver cancer. Worldwide, there are more than 700000 new cases of liver cancer every year, 55% of which are concentrated in China, which is the fourth most common malignant tumor and the third leading cause of death in China. More importantly, the onset of liver cancer is hidden, and 70% to 80% of patients with liver cancer are in the middle and advanced stage when they are first diagnosed, so they lose the opportunity for surgical treatment. Therefore, liver cancer seriously affects the life and health of the people. For these unresectable middle and advanced liver cancer, that is, Barcelona stage (barcelona clinic liver cancer,BCLC) stage C, BCLC and the European Association for the study of liver Diseases ((European Association for the Study of Liver Diseases)) recommended transarterial chemoembolization (transarterial chemoembolization,TACE) and systematic treatment, respectively. However, a number of clinical studies have shown that the prognosis of patients with advanced liver cancer who underwent surgical resection is significantly better than that of TACE or systemic therapy alone. Therefore, how to convert unresectable liver cancer into resectable liver cancer has always been a hot issue in clinical research.

Hepatectomy is to reduce the tumor load and tumor stage through some or several treatments, so that unresectable liver cancer can become resectable liver cancer and tumor resection. There are two purposes of translational therapy: one is that translational therapy can reduce tumor size, reduce tumor stage and improve its biological characteristics; the other is that translational therapy can select tumors with good biological characteristics. In 1977, Shafer et al reported that a single unresectable hepatoblastoma was successfully resected after radiotherapy and chemotherapy, and first mentioned the concept of liver cancer transformation therapy. Subsequently, sitzmann, Tang and fan reported the use of 131I or 90Y labeled anti ferritin antibody, TACE and TACE in the treatment of unresectable liver cancer. Finally, 8% to 18% of HCC patients underwent transformation resection. To be sure, the combination of multiple ways of transformation therapy can improve the success rate of transformation and prolong the survival of patients. But these studies are retrospective, the sample size is small, and the treatment plan is lack of unity. In addition, with the continuous emergence of targeted drugs and immune checkpoint blocking therapy (such as programmed death receptor-1, PD-1), the treatment mode of liver cancer has changed, and the success rate of transformation and resection may also be improved. Therefore, a prospective clinical study is urgently needed to explore the safety and effectiveness of hepatectomy in the new era of molecular targeted drugs and immunotherapy.

The treatment of liver cancer transformation includes local treatment and systemic therapy. The former includes TACE, transcatheter embolization, radiofrequency ablation, percutaneous alcohol injection, etc., among which TACE is the most commonly used local treatment. Fan and other scholars analyzed 65 patients with TACE after operation for liver cancer: the diameter of median tumor decreased from 9.9cm to 3.7cm, 35.9% (14/39) patients recovered AFP level, and the 1-year, 3-year and 5-year survival rate of patients were 80%, 65% and 56%, respectively. However, the pathological findings showed that 83.1% (54/65) of the tumors still failed to complete necrosis. Obviously, TACE is difficult to achieve complete necrosis of tumor as a non radical treatment. Moreover, the lack of 4 blood damage caused by TACE can induce the up regulation of related molecules (such as vascular endothelial growth factor (VEGF) which can promote the growth, invasion and metastasis of tumor. Therefore, TACE combined with antiangiogenic drugs can theoretically inhibit the angiogenesis and tumor growth induced by TACE, and TACE can reduce tumor effect or permit sensitization of antiangiogenic drugs. Solafeni and lumbotinib are first-line systemic therapy drugs for advanced liver cancer patients approved by FDA and CFDA. As a multi-target receptor tyrosine kinase inhibitor (TKI), they mainly inhibit VEGF receptor-1,2,3, FGF receptor-1,2,3,4, PDGFR α, RET and kit, thus inhibiting the proliferation of tumor cells, inducing apoptosis and playing an anti angiogenesis role. However, compared with solafeni, the binding of lumbotini with target molecules has stronger affinity. Based on an open label, multicenter, phase III non inferior effect clinical study, the results showed that the median survival time (13.6 months vs. 12.3 months) of the patients with liver cancer was the same as that of solafeni group, but the progression time (9.2 months vs. 3.6 months) and objective remission rate (24.1% vs. 9.2%) were better than those in the solafeni group. Therefore, TACE combined with lumbotinib may have better clinical outcomes.

Immune checkpoint blocking therapy may enhance the immune response induced by local treatment. TACE and other local treatment can make the body produce immune response. Local treatment leads to tumor cell death, apoptosis (non-cell necrosis) induces specific immunity of tumor, such as the release of calcium net protein and other endoplasmin on the cell surface, ATP secretion during the apoptosis and foaming stage, and the release of high mobility group box associated with cell death of non-histone chromatin group 1 1. HMGB1) promotes the collection, activation and entry of dendritic cells into the tumor microenvironment. The tumor antigen of tumor cells is phagocyted and the best antigen is presented to T cells. This process is called immunogenic cell death (ICD). Adriamycin (epirubicin, doxorubicin) as the most commonly used chemotherapeutic agent of TACE can enhance the immunogenicity of ICD. Therefore, TACE has been shown to promote ICD and induce tumor associated antigen-specific reactions. Ni Quanfa et al. Found that the levels of CD3 +, CD4 +, CD4 + / CD8 + increased significantly at 3 and 4 weeks after TACE treatment. Liao Juan and other researchers found that TACE can correct the low immune function of patients with HCC and make them partially recover. Kazumasa hiroishi and others studied 20 patients with HCC receiving TACE and RFA respectively. 80% of patients produced tumor specific antibody and cd8+ immune response one month later. Lakshmana ayaru et al. Found that APF specific CD4 + T cells increased after HCC embolization. Immune checkpoint blockade refers to blocking the inhibitory receptors or ligands on the surface of T cells, such as PD-1 / PD-L1, CTLA4 and Vista, to partially reverse T cell failure and improve tumor T cell response. This innovative treatment has been verified in a variety of solid tumors. Sangro et al. Showed that local treatment combined with immune checkpoint blocking therapy is safe and effective in patients with liver cancer. Moreover, TACE combined with immune checkpoint blocking therapy can further enhance the anti-tumor immunity without overlapping toxicity. Subsequently, a large number of clinical trials, such as nct03572582, nct03383458, nct03397654, were carried out worldwide to evaluate the efficacy of local treatment combined with immune checkpoint blocking therapy in patients with liver cancer.

In conclusion, current studies have shown that transformation therapy can benefit patients with unresectable HCC, but there are still some problems, such as low success rate of transformation, limited treatment options and so on. However, the new first-line drug for liver cancer is synergistic with TACE, and immune checkpoint blocking therapy may enhance the immune response induced by TACE. Therefore, this study is to compare the success rate of TACE combined with lenvastinib and sindilimab in the treatment of advanced unresectable liver cancer, and to explore the feasibility of the combined regimen in the treatment of liver cancer.

The clinical trial was monitored and audited by Ethics Committee on biological research, West China Hospital of Sichuan University.We will arrange special personnel in charge to compare the research data with the electronic medical records of West China hospital to ensure data consistency.The indexes we included refer to World Health Organization drug dictionary, MedDRA.The patients included in this clinical study were unresectable hepatocellular carcinoma patients. According to the existing guidelines, local treatment (such as TACE) and / or systemic treatment (lenvastinib) were the preferred treatment. Other treatment options include other targeted drugs (sorafenib), radiotherapy, chemotherapy and traditional Chinese medicine.In addition to regular follow-up and recording of the above examination results, patients undergoing transformation resection also need to be followed up and recorded in detail the postoperative combined treatment (radiotherapy, chemotherapy, immunotherapy, traditional Chinese medicine treatment) and combined medication (anti hepatitis B virus drugs, interferon, thymosin, other immunity enhancing drugs, Chinese patent medicine) and so on The starting and ending date, dosage and frequency of medication were analyzed. For the patients with failure of transformation resection, whether in the experimental group or the control group, they were still followed up every 3-4 months until the end of the event or the end of the trial. During each follow-up, the subjects, their family members or local doctors were asked by telephone or on-site visit. The window was opened for 10 days to collect the relapse / death (relapse / death date and cause of death) and the combined treatment information after the study treatment. Each survival follow-up should be recorded in the follow-up table.71 people are expected to be included in the experimental group and the control group, and the lost follow-up rate is less than 20%。Whether it is related to the research measures or not, any adverse medical event that is related to any medical measure in the study, unexpected, and adverse medical events are adverse events (AE). All observed or actively provided AE, whether caused by any study group or research measure, shall be recorded on AE page of pathological report. Serious adverse events shall be reported to ethics and relevant health administrative departments within 24 hours, and timely diagnosis and treatment shall be given.

The main researchers organize relevant training to ensure the research specifications are carried out, the filling of case report form or research record form and other reports follow GCP principles and research programs. TACE treatment for all patients is the responsibility and implementation of Professor luwusheng, liver surgery. The patients purchased the drug by themselves, and the patients actively recorded the drug taking cards during the drug administration. The silimab is kept by GCP center and is provided to patients free of charge. All data and treatment must be verifiable: in order to ensure the reliability of the study data, all observations and findings should be verifiable. Quality control will be used in every stage of the study to ensure the reliability of all data and the accuracy of the research procedure. The main investigator should ensure that the researchers comply with the test plan, confirm the accuracy of the data and the completeness of the record report, and ensure that informed consent from all subjects is obtained before the study begins. Any breach or deviation shall be reported to the ethics committee in a timely manner. If necessary, the research team will formulate standard operation procedures, and implement quality control procedures in all links of research and data processing to ensure the specification and reliability of research implementation and data operation.The clinical research will formulate corresponding data security monitoring plan according to the risk. All adverse events were recorded in detail, properly handled and tracked until they were properly resolved or stable, and serious adverse events and unexpected events were timely reported to ethics committee, competent department, sponsor and drug regulatory department according to regulations; main researchers conducted cumulative review on all adverse events on a regular basis, and convened a meeting of researchers to assess the risk of the study when necessary And benefit from it; Statistical analysis was performed by a specially assigned person (blind method). Statistical software SPSS V16.0 was used to analyze the data. The continuous variables were analyzed by unpaired Student's t test or Mann Whitney U test. The counting data were analyzed by chi square or Fisher's exact test. P < 0.05 was considered to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

-(1) 18 years old ≤ age ≤ 70 years old, no gender limit; (2) HCC patients who are in strict compliance with the clinical diagnostic criteria of the "Guidelines for the Diagnosis and Treatment of Hepatocellular Carcinoma (2019 Edition) or confirmed by histopathology or cytology; (3) Have not received any systemic treatment for HCC in the past. (4) ECOG PS score 0-1; (5) Child-Pugh liver function rating AB; (6) Patients with BCLC stage B and C liver cancer; or stage A patients without sufficient remaining liver volume (no cirrhosis liver: SFLVR<30%; cirrhosis liver: SFLVR<40%); (7) According to the evaluation criteria for the efficacy of solid tumors (mRECIST), there is at least one imaging measurable lesion; (8) If the patient is HBsAg positive, HBV-DNA will be less than 2000 IU/ml (10000 copies/ml) during PD-1antibody treatment; (9) The function of major organs is normal, that is, it meets the following standards:

1. . Sufficient bone marrow function, defined as: Absolute neutrophil count (ANC greater than or equal to 1.5×10^9 per liter (/L); hemoglobin (Hb greater than or equal to 8.5 grams per deciliter (g/dL); platelet count greater than or equal to 75×10^9/L).
2. . Sufficient liver function, defined as: Aspartate aminotransferase (AST), alkaline phosphatase (ALP) and alanine aminotransferase (ALT) are less than or equal to 5 ULN.
3. . Sufficient coagulation function, defined as the International Normalized Ratio (INR) less than or equal to 2.3.
4. . Sufficient renal function is defined as a creatinine clearance rate greater than 40 milliliters per minute (mL/min), calculated according to Cockcroft and Gault formulas.
5. . Sufficient pancreatic function, defined as amylase and lipase≤1.5×ULN.
6. . Normal thyroid function is defined as thyroid stimulating hormone (TSH) within the normal range. If the baseline TSH is outside the normal range, subjects whose total T3 (or FT3) and FT4 are within the normal range can also be included in the group; (10) Use up to 3 antihypertensive drugs to adequately control blood pressure (BP), defined as BP <= 150/90 mmHg at the time of screening, and there is no change in antihypertensive treatment within 1 week before cycle 1/day 1. .

(11) The patient is expected to survive more than 3 months. (12) No pregnancy or pregnancy plans. (13) The subjects voluntarily joined the study and signed an informed consent form, with good compliance and cooperation with follow-up.

Exclusion Criteria:

* (1) Extrahepatic metastasis of primary liver cancer; (2) Diffuse liver cancer, intrahepatic tumor burden ≥50%; portal vein tumor thrombus (superior mesenteric vein tumor thrombus, type IV), inferior vena cava tumor thrombus; (3) Contraindications of TACE and epirubicin; (4) Those who have participated in other clinical trial drugs within 4 weeks; (5) Those who are known to be allergic to the ingredients of lenvatinib; (6) Those who are known to be allergic to the active ingredients or excipients of Sintilizumab; (7) A history of liver resection, liver transplantation, interventional therapy, and other malignant tumors; (8) Women who are pregnant or breast-feeding; those with fertility who are unwilling or unable to take effective contraceptive measures; (9) Patients with grade II or higher myocardial ischemia or myocardial infarction, poorly controlled arrhythmia (including QTc interval ≥470 ms); according to NYHA standards, grade III to IV cardiac insufficiency, or cardiac color Doppler ultrasound examination suggests left ventricular ejaculation Blood score LVEF<50%; (10) Abnormal coagulation function (INR>1.5 or prothrombin time (PT)>ULN+4 seconds or APTT>1.5 ULN), have bleeding tendency or are receiving thrombolytic or anticoagulant therapy; (11) Have a mental illness or a history of psychotropic drug abuse; (12) Combined with HIV-infected patients; (13) Known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation; (14) Patients with active infection; (15) Patients with poor compliance such as floating population; (16) Have received the following therapies in the past: anti-PD-1, anti-PD-L1 or anti-PD-L2 drugs or for another stimulating or synergistic inhibition of T cell receptors (for example, CTLA-4, OX-40, CD137) medicine; (17) An active autoimmune disease that requires systemic treatment (such as the use of disease-relieving drugs, glucocorticoids, or immunosuppressive agents) occurred within 2 years before the first administration. Replacement therapies (such as thyroxine, insulin, or physiological glucocorticoids for adrenal or pituitary insufficiency, etc.) are not considered systemic treatments; (18) Are receiving systemic glucocorticoid therapy (excluding nasal spray, inhalation or other local glucocorticoids) or any other form of immunosuppressive therapy within 7 days before the first administration of the study; Note: physiological doses are allowed Glucocorticoids (≤10 mg/day prednisone or equivalent); (19) There is clinically uncontrollable pleural effusion/abdominal effusion (patients who do not need to drain the effusion or stop drainage for 3 days without a significant increase in effusion can be included in the group); (20) Acute or chronic active hepatitis B or C infection, HBV DNA ≥ 200000IU/ml or 106 copies/ml when Sintilimab is treated; hepatitis C virus HCV RNA ≥ 103 copies/ml; Hepatitis B surface anti-(HbsAg) and anti-HCV antibodies are positive at the same time.

  (21) Live vaccine has been vaccinated within 30 days before the first dose (cycle 1, day 1); Note: It is allowed to receive the inactivated virus vaccine for seasonal influenza injection within 30 days before the first dose; but it is not allowed to receive intranasal vaccine Medicated live attenuated influenza vaccine.

  (22) The researcher believes that it is not suitable for inclusion in the group.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Conversion resection rate | 48 weeks
  ratio of conversion resection patients / enrolled patients

SECONDARY OUTCOMES:
Objective Response Rate | 48 weeks
  It was defined as the percentage of patients with complete response (CR) and partial response (PR) in all patients, and the treatment response was based on the modified response evaluation criteria in solid tumors (mrecist)
PFS | 96 weeks
  It was defined as the time from successful hepatectomy to recurrence. Patients who withdraw or lose follow-up will be treated as deletion.
OS | 96 weeks
  It was defined as the time from the beginning of treatment to death from any cause throughout the trial. Patients who dropped out or lost follow-up will be treated as deletion, and the known last survival date will be regarded as the last survival time. Patients who survived at the end of the study will also be treated as deletions, and the last known date of survival will be taken as the final survival time

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided
On March 20, 2025, ResMan (www.medresman.org) etc.